CLINICAL TRIAL: NCT03503305
Title: Healing Osteoarthritic Joints in the Wrist With Adult Adipose Derived Regenerative Cells
Brief Title: Healing Osteoarthritic Joints in the Wrist With Adult ADRCs
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: InGeneron, Inc. (Industry)
Collaborators: Sanford Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OAW-001
Record Dates: First submitted 2018-04-05; First posted 2018-04-19 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Osteoarthritis of the Wrist
Keywords: Adipose-derived stem cells; osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: It is a double-blinded trial in which the subjects, investigator and radiologists are blinded to treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Adipose Derived Regenerative Cell group (Experimental): Subjects in the treated group will receive an Adipose derived regenerative cells (ADRCs) injection into the wrist using a fluoroscopic-guided injection .
  Interventions: Device: adipose-derived stem cell injection
- Corticosteroid group (Active Comparator): Subjects in the active control group will receive a corticosteroid injection into the wrist using a fluoroscopic-guided injection.
  Interventions: Drug: Corticosteroid injection

INTERVENTIONS:
Device: adipose-derived stem cell injection — 5 ml injection of adipose derived stem cells
  Arms: Adipose Derived Regenerative Cell group
Drug: Corticosteroid injection — 5 ml injection of corticosteroid
  Arms: Corticosteroid group

SUMMARY:
This is a prospective, randomized, double-blinded, active controlled, single site safety and efficacy study in subjects suffering from chronic wrist osteoarthritis comparing a single ADRC injection generated with the Transpose® RT system into the wrist.

DETAILED DESCRIPTION:
The focus of this study is to investigate the therapeutic benefit of autologous adipose-derived regenerative cells in patients with wrist arthritis. The hypothesis of this trial is that the use of adult-adipose derived regenerative cells as a treatment of wrist arthritis will induce healing and decrease pain compared to the control group. With adult-adipose derived regenerative cell administration, the medical practitioner would anticipate a reduction in inflammation, acceleration in healing, decreased pain in patients post procedure, and increased function and strength in the affected wrist. Currently, no clinical studies have been constructed to determine the efficacy of ADRCs in wrist arthritis patients.

Subjects will fall into two categories: treatment group (20) and control group (20 subjects). The treatment group will undergo a small liposuction procedure and receive wrist osteoarthritis treatment with an ultrasound-guided injection of 5 ml adipose-derived stem cells (ADSCs) into the wrist. The control group will receive a 5 ml cortisone injection into the wrist.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ages: 18 - 75.
2. Clinical symptoms consistent with wrist osteoarthritis.
3. Diagnosed with wrist osteoarthritis on radiographs.
4. The ability of subjects to give appropriate consent or have a legally authorized representative available.

Exclusion Criteria:

1. Subjects who have a documented history or presence of inflammatory arthritis, rheumatoid arthritis, severe osteoporosis, sepsis and chondrocalcinosis in the wrist
2. Subjects who have a documented diagnosis of carpal tunnel syndrome.
3. Insufficient amount of subcutaneous tissue to allow recovery of 100ml of lipoaspirate
4. History of systemic malignant or local neoplasms on affected limb within last 5 years
5. Subject is receiving immunosuppressant therapy or has known immunosuppressive or severe autoimmune disease that requires chronic immunosuppressive therapy (e.g., human immunodeficiency virus, systemic lupus erythematosus, etc.)
6. Subjects who have received a corticosteroid injection in the treatment site
7. Subjects on an active regimen of chemotherapy
8. Allergy to sodium citrate of any "caine" type of local anesthetic
9. Subjects pregnant or breast feeding
10. Subject is in the opinion of the Investigator or designee, unable to comply with the requirements of the study protocol or is unsuitable for the study for any reason. This includes completion of patient reported outcome instruments
11. Subjects who have document allergy to radiographic guidance agents.
12. Subject is currently participating in another clinical trial that has not yet completed its primary endpoint
13. History of tobacco use within the last 3 months
14. Subjects with documented with a history of alcohol or drug abuse
15. Subjects who have a documented history of HIV, Hepatitis B, and Hepatitis C
16. Subject is part of a vulnerable population who, in the judgment of the investigator, is unable to give Informed Consent for reasons of incapacity, immaturity, adverse personal circumstances or lack of autonomy. This may include: Individuals with mental disability, persons in nursing homes, children, impoverished persons, persons in emergency situations, homeless persons, nomads, refugees, and those incapable of giving informed consent. Vulnerable populations also may include members of a group with a hierarchical structure such as university students, subordinate hospital and laboratory personnel, employees of the Sponsor, members of the armed forces, and persons kept in detention.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-11-21 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Safety - Incidence of Treatment-Emergent Adverse Events | 12 months
  Subjects will be monitored for adverse events

SECONDARY OUTCOMES:
Efficacy - Change in Pain Scores on the Visual Analog Scale (VAS)-pain Scale at All Follow-up Visits | 3, 6 and 12 months
  Patient outcomes for pain will be recorded (line from 0: no pain to 100:worst pain)
Efficacy - Change in Function Scores on the PROMIS at All Follow-up Visits | 3, 6 and 12 months
  Patient outcomes for function will be recorded (line from 0:unable to do to 100: without any difficulty)
Efficacy - Change in Function Scores on the QuickDASH at All Follow-up | 3, 6 and 12 months
  Patient outcomes for function will be recorded (line from 0:no difficulty to 100:unable)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Sanford USD Medical Center, Sioux Falls, South Dakota
  - HD Research, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gimble JM, Katz AJ, Bunnell BA. Adipose-derived stem cells for regenerative medicine. Circ Res. 2007 May 11;100(9):1249-60. doi: 10.1161/01.RES.0000265074.83288.09. PMID 17495232
- [Background] ter Huurne M, Schelbergen R, Blattes R, Blom A, de Munter W, Grevers LC, Jeanson J, Noel D, Casteilla L, Jorgensen C, van den Berg W, van Lent PL. Antiinflammatory and chondroprotective effects of intraarticular injection of adipose-derived stem cells in experimental osteoarthritis. Arthritis Rheum. 2012 Nov;64(11):3604-13. doi: 10.1002/art.34626. PMID 22961401
- [Background] Jo CH, Lee YG, Shin WH, Kim H, Chai JW, Jeong EC, Kim JE, Shim H, Shin JS, Shin IS, Ra JC, Oh S, Yoon KS. Intra-articular injection of mesenchymal stem cells for the treatment of osteoarthritis of the knee: a proof-of-concept clinical trial. Stem Cells. 2014 May;32(5):1254-66. doi: 10.1002/stem.1634. PMID 24449146